CLINICAL TRIAL: NCT06343558
Title: Gait and Balance Impairment in Rare and Very Rare Neurological Diseases
Acronym: GALVANISE
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: IRCCS Istituto Neurologico Carlo Besta (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24C302
Record Dates: First submitted 2024-03-08; First posted 2024-04-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Parkinson Disease; Peripheral Neuropathy; Rare Diseases; Healthy; Healthy Aging
Keywords: Rare neurological diseases; Very rare neurological diseases; Undiagnosed neurological diseases; Upright stance; Balance; Risk of falling; Gait analysis; Posturography
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease; Peripheral Nervous System Diseases; Rare Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy controls
  Interventions: Other: Questionnaires, clinical scales and instrumental tests
- Parkinson's disease patients
  Interventions: Other: Questionnaires, clinical scales and instrumental tests
- Multiple sclerosis patients
  Interventions: Other: Questionnaires, clinical scales and instrumental tests
- Peripheral neuropathies of the lower limbs
  Interventions: Other: Questionnaires, clinical scales and instrumental tests
- Rare and ultrarare neurological diseases
  Interventions: Other: Questionnaires, clinical scales and instrumental tests

INTERVENTIONS:
Other: Questionnaires, clinical scales and instrumental tests — Questionnaires, clinical scales and instrumental tests to collect a wide range of balance and gait measures.

SUMMARY:
Rare and very rare neurological diseases primarily or exclusively affect the nervous system with a prevalence of < 5 out of 10'000 and 100'000 people, respectively. Besides these, there are undiagnosed neurological diseases: neurological conditions without a diagnosis after completing a full diagnostic examination.

Rare, very rare, and undiagnosed neurological diseases are complicated and progressive and often cause variegated motor signs, impairments, and syndromes.

Balance and gait are frequently affected in these conditions, already at the clinical examination. These balance and gait impairments limit activities and cause an increased risk of falling. Falls can eventually result in injuries, even severe.

There are only a few studies about these diseases, likely because of their rarity. Hence, the clinical presentation and the course of rare and very rare diseases are poorly known or even unknown. Essential information for these conditions' diagnosis, prognosis, treatment and rehabilitation is missing.

MaNeNeND is an observational study underway at the Fondazione IRCCS Istituto Neurologico "Carlo Besta" (Milano) aimed at detailing the clinical and biological features of very rare and undiagnosed neurological diseases.

Research questions:

1. Do patients with rare (Ra), very rare (V) and undiagnosed (U) neurological diseases suffer a balance and gait impairment?
2. Is there a correlation between the clinical and instrumental severity of the balance and gait impairment in RaVU neurological diseases?
3. Are instrumental measures more sensitive in detecting balance and gait impairments in patients affected by a RaVU neurological disease than the clinical measures?
4. Do the balance and gait impairments in RaVU neurological diseases worsen in time?

The current project aims at diagnosing, quantifying and detailing the balance and gait impairment in rare, very rare and undiagnosed neurological diseases.

To this aim, questionnaires, clinical scales and instrumental tests will be administered to these patients to collect a wide range of balance and gait measures.

These measures will also integrate those collected with MaNeNeND to provide a more detailed description of patients with rare, very rare and diagnosed neurological diseases.

Participants will complete two questionnaires: the Dizziness Handicap Inventory - short form (DHI-sf, an ordinal score of self-perceived balance) and the Modified Fatigue Impact Scale (MFIS, an ordinal score of self-perceived fatigue).

Moreover, a clinician will administer the Mini Balance Evaluation Systems Test (Mini-BESTest, an ordinal score of balance), the 10 m walking test (for measuring the gait speed and other gait parameters) and the Timed Up and Go test (an instrumental measure of mobility and balance). Walking and the Timed Up and Go tests will be recorded with a trunk-worn inertial measurement unit.

Finally, participants will be asked to complete an instrumental upright stance and gait assessment, the first consisting of standing on posturographic plates and the second of walking on a treadmill equipped with force sensors. When walking on the treadmill, an optoelectronic system will also record the position in time of limbs and trunk.

The quantification of the severity of the balance and gait impairment of the patients suffering a rare, very rare or undiagnosed neurological disease will highlight these persons' therapeutic and rehabilitative needs.

Comparing the balance and gait impairment of rare, very rare and undiagnosed diseases with those of multiple sclerosis, Parkinson's disease and peripheral neuropathy will highlight if the formers' balance and gait impairment has unique characteristics that could help ease the diagnosis of these uncommon conditions.

The longitudinal measurements on rare, very rare and undiagnosed diseases will be paramount to identifying prognostic factors.

In addition, the data collected in the current study will be crucial for future studies, for example, for estimating the sample size in clinical trials.

ELIGIBILITY:
Inclusion criteria

* Multiple sclerosis, Parkinson's disease, peripheral neuropathy of the lower limbs or rare or ultrarare neurological disease (e.g. la Cerebellar Ataxia with Neuropathy and Vestibular Areflexia Syndrome - CANVAS, ORPHAcode: 504476; Wilson's disease, ORPHAcode: 905)
* undiagnosed neurological disease, i.e. a neurological disease that remains unknown after a full diagnostic assessment;
* age > 18 years;
* ability to stand upright with no assistance and no assistive device for > 30 seconds;
* ability to walk without assistance and with no assistive device for > 50 m;
* ability to give their informed consent.

Exclusion criteria

* pregnancy or breastfeeding
* any other medical conditions affecting by itself balance and gait (e.g. lower limb amputation, hemiparesis due to a stroke)
* major orthopaedic surgery (e.g. hip or knee replacement).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with a balance and gait impairment secondary to multiple sclerosis, Parkinson's disease, peripheral neuropathy of the lower limbs, a rare, ultrarare or undiagnosed neurological disease.
  A group of age-matched controls will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Balance (Mini-BESTest) | At enrollment
  Mini Balance Evaluation Systems Test (Mini-BESTest, an ordinal score of balance)
Balance (Timed Up and Go test) | At enrollment
  Timed Up and Go test instrumented with inertial sensors
Gait speed | At enrollment
  10 m walking test
Gait analysis - kinematic - stride length | At enrollment
  Stride length, right step length and left step length
Gait analysis - kinematic - duration | At enrollment
  Stride duration, right and left step duration
Gait analysis - kinematic - width of the base of support | At enrollment
  Width of the base of support
Gait analysis - kinematic - dorsal ankle angle | At enrollment
  Dorsal ankle angle
Gait analysis - dynamic - reaction force | At enrollment
  Anterior-posterior, mediolateral and vertical reaction force
Gait analysis - dynamic - ankle power | At enrollment
  Right and left ankle power
Gait analysis - dynamic - energy | At enrollment
  Potential and kinetic energy of the body centre of mass
Posturography - static - centre of pressure position | At enrollment
  Centre of pressure position while standing
Posturography - static - centre of mass position | At enrollment
  Centre of mass position while standing
Posturography - dynamic - centre of pressure position | At enrollment
  Centre of pressure position after base of support perturbations
Posturography - dynamic - centre of mass position | At enrollment
  Centre of mass position after base of support perturbations

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Istituto Auxologico Italiano, Milan, Milan
  - IRCCS Istituto Neurologico Carlo Besta, Milan

IPD SHARING:
Plan to Share IPD: No
The database will be made available upon request on Zenodo.

REFERENCES:
- [Background] Reinhard C, Bachoud-Levi AC, Baumer T, Bertini E, Brunelle A, Buizer AI, Federico A, Gasser T, Groeschel S, Hermanns S, Klockgether T, Krageloh-Mann I, Landwehrmeyer GB, Leber I, Macaya A, Mariotti C, Meissner WG, Molnar MJ, Nonnekes J, Ortigoza Escobar JD, Perez Duenas B, Renna Linton L, Schols L, Schuele R, Tijssen MAJ, Vandenberghe R, Volkmer A, Wolf NI, Graessner H. The European Reference Network for Rare Neurological Diseases. Front Neurol. 2021 Jan 14;11:616569. doi: 10.3389/fneur.2020.616569. eCollection 2020. PMID 33519696
- [Background] The Lancet Neurology. Rare neurological diseases: a united approach is needed. Lancet Neurol. 2011 Feb;10(2):109. doi: 10.1016/S1474-4422(11)70001-1. No abstract available. PMID 21256450
- [Background] Ganz DA, Bao Y, Shekelle PG, Rubenstein LZ. Will my patient fall? JAMA. 2007 Jan 3;297(1):77-86. doi: 10.1001/jama.297.1.77. PMID 17200478
- [Background] Vieira ER, Palmer RC, Chaves PH. Prevention of falls in older people living in the community. BMJ. 2016 Apr 28;353:i1419. doi: 10.1136/bmj.i1419. No abstract available. PMID 27125497
- [Background] Caronni A, Sterpi I, Antoniotti P, Aristidou E, Nicolaci F, Picardi M, Pintavalle G, Redaelli V, Achille G, Sciume L, Corbo M. Criterion validity of the instrumented Timed Up and Go test: A partial least square regression study. Gait Posture. 2018 Mar;61:287-293. doi: 10.1016/j.gaitpost.2018.01.015. Epub 2018 Jan 31. PMID 29413799
- [Background] Picardi M, Redaelli V, Antoniotti P, Pintavalle G, Aristidou E, Sterpi I, Meloni M, Corbo M, Caronni A. Turning and sit-to-walk measures from the instrumented Timed Up and Go test return valid and responsive measures of dynamic balance in Parkinson's disease. Clin Biomech (Bristol). 2020 Dec;80:105177. doi: 10.1016/j.clinbiomech.2020.105177. Epub 2020 Sep 18. PMID 32979787
- [Background] Caronni A, Gervasoni E, Ferrarin M, Anastasi D, Brichetto G, Confalonieri P, Di Giovanni R, Prosperini L, Tacchino A, Solaro C, Rovaris M, Cattaneo D, Carpinella I. Local Dynamic Stability of Gait in People With Early Multiple Sclerosis and No-to-Mild Neurological Impairment. IEEE Trans Neural Syst Rehabil Eng. 2020 Jun;28(6):1389-1396. doi: 10.1109/TNSRE.2020.2991636. Epub 2020 Apr 30. PMID 32356754
- [Background] Scarano S, Sansone VA, Ferrari Aggradi CR, Carraro E, Tesio L, Amadei M, Rota V, Zanolini A, Caronni A. Balance impairment in myotonic dystrophy type 1: Dynamic posturography suggests the coexistence of a proprioceptive and vestibular deficit. Front Hum Neurosci. 2022 Jul 28;16:925299. doi: 10.3389/fnhum.2022.925299. eCollection 2022. PMID 35967003
- [Background] Scarano S, Rota V, Tesio L, Perucca L, Robecchi Majnardi A, Caronni A. Balance Impairment in Fahr's Disease: Mixed Signs of Parkinsonism and Cerebellar Disorder. A Case Study. Front Hum Neurosci. 2022 Mar 9;16:832170. doi: 10.3389/fnhum.2022.832170. eCollection 2022. PMID 35355583